CLINICAL TRIAL: NCT01001676
Title: Local Delivery of Paclitaxel for Prevention of Restenosis in Hemodialysis Access
Brief Title: Restenosis Following Paclitaxel Eluting Balloon Angioplasty of Hemodialysis Access Stenosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ktt1
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2012-01

CONDITIONS: Renal Failure
Keywords: renal failure; Restenosis; Dialysis access; Paclitaxel; Angioplasty; Intimal hyperplasia
MeSH Terms: conditions — Renal Insufficiency | interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Balloon Angioplasty (Active Comparator)
  Interventions: Device: Percutaneous Transluminal Angioplasty (PTA)
- Drug Eluting Balloon Angioplasty (Experimental)
  Interventions: Device: Paclitaxel Eluting Balloon Angioplasty

INTERVENTIONS:
Device: Percutaneous Transluminal Angioplasty (PTA) — Angioplasty with the use of Conventional balloon
  Arms: Conventional Balloon Angioplasty
Device: Paclitaxel Eluting Balloon Angioplasty — Angioplasty with the use of paclitaxel eluting balloon
  Other Names: Passeo-18 Lux (Biotronik)
  Arms: Drug Eluting Balloon Angioplasty

SUMMARY:
Introduction: Narrowing of the draining vein occurs in >50% of hemodialysis fistula and left untreated will lead to loss of access. The narrowing is due to excessive growth of tissue in the vessel wall (intimal hyperplasia). The standard treatment is balloon dilatation. However, narrowing will inevitably recur in 2-3 months hence requiring further dilatation. Intimal hyperplasia also occurs in the heart and leg circulation. The drug paclitaxel has been used with great success in preventing intimal hyperplasia in these vessels following balloon dilatation. Administer locally, paclitaxel inhibits excess tissue growth in the vessel wall. The investigators believe that this drug will have similar effect in hemodialysis access..

Objective: To assess the effect of paclitaxel in hemodialysis access with narrowing. Paclitaxel is delivered by a paclitaxel-coated balloon. This balloon dilates the narrow segment and simultaneously delivers paclitaxel to the vessel wall.

Methodology: Patients with narrowed hemodialysis access are dilated with the paclitaxel-coated balloon or conventional balloon in randomized manner. The patency of the two groups are evaluated and compared at 6 months follow-up.

Potential benefit: Decrease number of balloon dilatations and hence hospital admissions, improve dialysis fistula function, and decrease overall economic cost.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis access located in the forearm or upper arm
* Patient with clinical or hemodynamic evidence of graft dysfunction
* Hemodialysis access is > 3 months old

Exclusion Criteria:

* Intervention of the vascular access circuit within the past 30 days
* Thrombosed/clotted access
* Evidence of systemic infection or a local infection associated with the graft
* Positive pregnancy test within 7 days before enrolment
* Patient is scheduled for a kidney transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Primary patency | at 6 months

SECONDARY OUTCOMES:
Transonic blood flows | monthly for up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kong Teng Tan, BCh MB, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada